CLINICAL TRIAL: NCT01172288
Title: Double-Blind, Placebo-Controlled Trial of N-acetylcysteine (NAC) for the Treatment of Children With Tourette Syndrome
Brief Title: N-acetylcysteine (NAC) for Children With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YCSC1004006637
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Tourettes Syndrome; Tic
Keywords: Tic disorders,; Tourette syndrome; Chronic Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tics; Tic Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): NAC was titrated up to a maximum dose of 2400 mg over the course of 2 weeks. Subjects were assigned 600 mg twice a day for weeks 1-2, and then were assigned 1200 mg twice a day for the remainder of the 12 week study.
  Interventions: Drug: N-Acetylcysteine (NAC)
- Placebo (Placebo Comparator): Placebo: Subjects were assigned to take two capsules twice a day for weeks 1-2, and then were assigned 4 capsules twice a day for the remainder of the 12 week study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — 1 600mg capsule twice a day for 2 weeks and then 2 600mg capsules twice a day for the remaining 10 weeks of the trial.
  Arms: N-Acetylcysteine
Drug: Placebo — 1 600mg Capsule twice a day for two weeks then 2 600mg capsules twice a day for the remaining 10 weeks of the study. Children receiving placebo will be offered the active intervention after the double-blind portion of the trial.
  Arms: Placebo

SUMMARY:
Tourette syndrome is a childhood-onset neuropsychiatric disorder characterized by multiple motor and vocal tics that last for at least a year in duration. Currently, there exist several effective pharmacological treatments for childhood tics including alpha-2 agonist medications (guanfacine and clonidine) and neuroleptics (antipsychotic) medications. These medications, however, have significant side-effects and are only partially efficacy in treating tics.

N-acetylcysteine (NAC) is a natural supplement that acts as an antioxidant and glutamate modulating agent. NAC has been used safely for decades in doses 20-40 times higher than in this trial as an antidote for acetaminophen overdose. The only side-effect commonly seen with NAC is nausea and this side-effect is seldom seen in the doses used in this trial.

NAC has recently been demonstrated to be effective in a double-blind, placebo-controlled trial in adults with trichotillomania (chronic hair pulling). Hairpulling is hypothesized to be closely related to tics because these conditions (1) have similar clinical characteristics -- both groups typically experience urges before engaging in pulling or tics, (2) neuroimaging studies suggest they involve similar brain circuits -- the basal ganglia, (3) the same pharmacological treatments (neuroleptics) may be effective for both conditions and (4) they tend to be inherited together in families. In other trials NAC has evidence of some efficacy in treating diverse psychiatric conditions such as bipolar depression, schizophrenia and cocaine dependence.

The investigators are conducting this trial to determine if NAC is an effective treatment for tics.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17 years.
* Primary diagnosis of Tourette syndrome or chronic tic disorder.
* Duration of tics greater than 1 year.
* Significant Current tic symptoms: Current YGTSS score greater than or equal to 22 with a TS diagnosis or greater than or equal to 14 with a chronic tic disorder.

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or mental retardation (IQ<70).
* Recent change (less than 4 weeks) in medications that have potential effects on tic severity (such as neuroleptic medications, dopamine agonists, alpha-2 agonists (guanfacine, clonidine or prazosin), SSRIs, clomipramine, naltrexone, lithium, psychostimulants, or anxiolytics). Medication change is defined to include dose changes or medication discontinuation.
* Recent change in behavioral treatment for Tourette syndrome or comorbid conditions (i.e. OCD) within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
* Asthma requiring medication use within the last 3 months
* Known hypersensitivity or previous anaphylactoid reaction to acetylcysteine or any components in its preparation
* Positive pregnancy test or drug screening test.
* Previous use of N-acetylcysteine (dose greater than 600mg for more than 2 weeks)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant JE, Odlaug BL, Kim SW. N-acetylcysteine, a glutamate modulator, in the treatment of trichotillomania: a double-blind, placebo-controlled study. Arch Gen Psychiatry. 2009 Jul;66(7):756-63. doi: 10.1001/archgenpsychiatry.2009.60. PMID 19581567
- [Background] Bloch MH, Leckman JF. Clinical course of Tourette syndrome. J Psychosom Res. 2009 Dec;67(6):497-501. doi: 10.1016/j.jpsychores.2009.09.002. PMID 19913654
- [Background] Berk M, Copolov DL, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Bush AI. N-acetyl cysteine for depressive symptoms in bipolar disorder--a double-blind randomized placebo-controlled trial. Biol Psychiatry. 2008 Sep 15;64(6):468-75. doi: 10.1016/j.biopsych.2008.04.022. Epub 2008 Jun 5. PMID 18534556
- [Background] Berk M, Copolov D, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Judd F, Katz F, Katz P, Ording-Jespersen S, Little J, Conus P, Cuenod M, Do KQ, Bush AI. N-acetyl cysteine as a glutathione precursor for schizophrenia--a double-blind, randomized, placebo-controlled trial. Biol Psychiatry. 2008 Sep 1;64(5):361-8. doi: 10.1016/j.biopsych.2008.03.004. Epub 2008 Apr 23. PMID 18436195
- [Background] Ng F, Berk M, Dean O, Bush AI. Oxidative stress in psychiatric disorders: evidence base and therapeutic implications. Int J Neuropsychopharmacol. 2008 Sep;11(6):851-76. doi: 10.1017/S1461145707008401. Epub 2008 Jan 21. PMID 18205981
- [Background] Singer HS, Morris C, Grados M. Glutamatergic modulatory therapy for Tourette syndrome. Med Hypotheses. 2010 May;74(5):862-7. doi: 10.1016/j.mehy.2009.11.028. Epub 2009 Dec 21. PMID 20022434
- [Result] Bloch MH, Panza KE, Yaffa A, Alvarenga PG, Jakubovski E, Mulqueen JM, Landeros-Weisenberger A, Leckman JF. N-Acetylcysteine in the Treatment of Pediatric Tourette Syndrome: Randomized, Double-Blind, Placebo-Controlled Add-On Trial. J Child Adolesc Psychopharmacol. 2016 May;26(4):327-34. doi: 10.1089/cap.2015.0109. Epub 2016 Mar 30. PMID 27027204
- See also: Yale Child Study Center TS/OCD Clinic — https://medicine.yale.edu/childstudy/ocd/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 17 | 14
Completed | 16 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (1.4) | 11.5 (2.8) | 11.9 (2.17)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 12 | 12 | 24
Age of onset [Mean (Standard Deviation); unit: years] | 6.8 (1.4) | 6.1 (2.4) | 6.4 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Tic Severity
Description: Yale Global Tic Severity Scale is a standard psychiatric measure that rates tics from 0 (no tics) to 100 (most severe tics).
  It separately rates motor tics and vocal tics in 5 subscales (number, frequency, intensity, complexity and interference) where the maximum severity score for motor tics is 25 and for vocal tics is 25. Giving us the Total Tic Severity Score maximum of 50.
  The additional Impairment Scale rates the degree of disability caused by the tics ranging from 0 (none) to 50 (severe). When these two scores are added we get the Yale Global Tic Severity Scale Score.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 17 | 14
units on a scale | 24.3 (7.9) | 21.3 (4.6)

2. Secondary Outcome: Improvement of Premonitory Urges
Description: Premonitory Urge for Tics Scale (PUTS). Items are rated on a scale of 1-4 from "least" to "most." A total score is calculated by summing the scores of all items. Nine is the minimum possible score. A score of 12.5-24.5 indicates medium intensity of premonitory urges for tics. A score of 25-30.5 indicates high intensity which may be associated with marked impairment. Scores 31 and above indicate extremely high intensity with probable severe impairment. A score of 36 is the maximum score possible.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 17 | 14
units on a scale | 24.7 (4.9) | 24.1 (4.8)

3. Secondary Outcome: Improvement in OCD Severity
Description: Childrens' Yale-Brown Obsessive-Compulsive Scale (CY-BOCS). 10-item scale. Each item is rated from 0-4. A sum total is calculated by adding items 1-10. 0-7: Subclinical. 8-15: Mild. 16-23: Moderate. 24-31: Severe. 32-40: Extreme.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 17 | 14
units on a scale | 4.4 (8.0) | 11.5 (9.8)

4. Secondary Outcome: Overall Improvement
Description: Clinical Global Impression - Improvement Scale (CGI-I). The CGI is a 7-point scare that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 17 | 14
units on a scale | 3.3 (1.1) | 3.4 (1.1)

5. Secondary Outcome: Number of Participants With Adverse Effects
Description: Number of participants with adverse events according to the Pediatric Adverse Events Rating Scale
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 17 | 14
participants
  Irritability | 0 | 0
  Sadness or depressed mood | 0 | 1
  Fatigue | 0 | 0
  Insomnia | 0 | 0
  Decreased appetite | 0 | 0
  Chest pain | 0 | 0
  Syncope | 0 | 0
  Stomach ache | 0 | 2
  Nausea | 0 | 3
  Vomiting | 0 | 0
  Headache | 1 | 1

ADVERSE EVENTS:
Time Frame: Every 4 weeks until the completion of the 12-week study
Description: Adverse events were systematically assessed with every assessment using the PAERS, unless they were brought to our attention by the subject between assessment periods.
Arm/Group | N-Acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 2/17 | 7/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=17) | Placebo (N=14)
Worsening of symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Subject dropped out of NAC arm because of worsening of tic symptoms.
Sadness or depressive mood (Psychiatric disorders) | 0 (0) | 1 (1)
Stomach Ache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No